CLINICAL TRIAL: NCT06514066
Title: Cannabidiol's Role in Dementia Management: Evaluating Cognitive, Quality of Life, and Well-being Outcomes in Malaysia
Brief Title: Cannabidiol's Role in Dementia Management
Acronym: MyC4D
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Pengajar Universiti Putra Malaysia (Other)
Collaborators: UPM Consultancy & Services Sdn. Bhd. (Unknown); Pure Life Collective Pte Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: CBDA102223
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Dementia, Vascular; Dementia, Mixed
MeSH Terms: conditions — Dementia, Vascular; Mixed Dementias | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Subjects will receive placebo for the first three months. After transitioning from the placebo, subjects will be titrated with 200 mg CBD for the first two weeks. Subsequent to this period, they will be administered 400 mg CBD for the remaining two and a half months.
  Interventions: Drug: Cannabidiol Oil
- Group B (Other): For the initial two weeks, subjects will be given 200 mg CBD. Following this titration period, they will receive 400 mg CBD for the remaining two and a half months. Then, subjects will receive placebo for the remaining of the study.
  Interventions: Drug: Cannabidiol Oil

INTERVENTIONS:
Drug: Cannabidiol Oil — The study intervention involves the administration of high purity Cannabidiol (CBD) in vegan soft gel capsule form. Dosing will range between 200 mg and 400 mg and will be administered twice daily. The CBD capsule is water-soluble to improve its bioavailability and absorption in the body.

SUMMARY:
This trial investigates the therapeutic benefits of cannabidiol (CBD) for Dementia patients in Malaysia. As dementia becomes increasingly prevalent worldwide, there's a pressing demand for impactful remedies. This research will delve into CBD's influence on cognitive functions, daily activities, mental health, and overall life quality of dementia sufferers. Utilizing a range of established assessment instruments, including the ADAS-COG subscale for cognitive effects, the NPI score for psychological well-being, and the QOLAD questionnaire for life quality, we aim to discern CBD's potential in ameliorating the conditions of those with dementia. This study's results could shape novel treatment methods and improved care for dementia patients, benefiting not just Malaysia but the world at large.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Participants (male and female) must be 50 years of age or older at the time of enrollment. This criterion is necessary to ensure that participants can legally provide informed consent for their participation.
2. Diagnosis: Participants must have a confirmed diagnosis of mild to severe dementia based on DSM-5 and Clinical Dementia Rating (CDR). Diagnosis should be confirmed by either neurologist, psychiatrist or geriatrician that attend the pattients.
3. Stability of Condition: Participants' disease status must be stable at the time of enrollment, as determined by the investigator. For example, seizure frequency for those with epilepsy should be consistent for a specified period (e.g., the past three months) before study entry.
4. Consent: The caregivers of the participants must provide written informed consent to participate in the study. The consent form must be read, understood, and signed by the caregivers before any study-specific procedures are performed.
5. Ability to Comply: Participants' caregivers must be willing and able to comply with all study procedures and requirements needed by the study. The caregivers must ensure that the participants has the ability to ingest oral medication, and they need to complete surveys on behalf of the participants on their phone, record log seizures (if applicable), and bring the patients to attend all necessary study visits.
6. Health Status: Participants must be in a health state, as determined by the investigator that will not put them at undue risk of harm from participating in the study or interfere with the study's ability to achieve its objectives.
7. Additional Criteria for Cancer Patients: Cancer patients must not be on any active chemotherapy and radiation treatment, as determined by the investigator.

The exact specifications of these criteria will be determined in consultation with Malaysian clinical experts and will be clearly defined in the study's protocol. These criteria are intended to ensure the study's results are valid, reliable, and applicable to the target population.

Exclusion Criteria:

1. Cannot fulfil all the requirement as above.
2. Substance Use: Active usage of substances/medications such as cocaine, opiates, benzodiazepines, barbiturates, amphetamines, morphine, methadone, methamphetamines, oxycodone, phencyclidine, tricyclic antidepressants, tetrahydrocannabinol, buprenorphine, methylenedioxymethamphetamine, propoxyphene.
3. Concurrent Treatments: Participants currently participating in another clinical trial or using other experimental treatments for their condition. Participants who have used any medication, dietary supplements (and/or grapefruit juice), or combination of medications and supplements known to alter the metabolism of, or interact with CBD (bupropion, rifampin, barbiturates, phenothiazines, cimetidine, etc.) 14 days prior to and during the duration of the study.
4. Significant Health Risks: Participants with significant cardiovascular, hepatic, renal, respiratory, or psychiatric disease, which, in the investigator's opinion, would place the participant at undue risk or interfere with the results of the study. History of impaired renal function or elevated liver enzymes at prescreening. The exclusionary lab values are: 3x nl AST/ALT, 1.5x bilirubin or eGFR less than 30 ml/min. Having present or past medical conditions, including a DSM-5 Axis I psychiatric disorder, history of cardiac disease, arrhythmias, neurological disease of central origin, head trauma, and seizures.
5. Hypersensitivity: Individuals with known hypersensitivity to CBD or any component of the study formulation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function: The Alzheimer's Disease Assessment Scale-Cognitive subscale (ADAS-COG) | 6 months
  To evaluate cognitive functions using the Alzheimer's Disease Assessment Scale-Cognitive subscale. The ADAS-COG consists of 11 tasks: Word Recall Task, Naming Objects and Fingers, Following Commands, Constructional Praxis, Ideational Praxis, Orientation, Word Recognition Task, Remembering Test Directions, Spoken Language, Comprehension, and Word-Finding Difficulty .
Psychological well-being/ assesses psycho-behavioral symptomatology (the Neuropsychiatric Inventory NPI scoring system) | 6 months
  To measure psychological well-being. The NPI evaluates neuropsychiatric symptoms through domains including delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition, irritability, apathy, and aberrant motor activity, each with 7-8 specific sub-questions assessing severity and frequency.
Sleep quality, latency, duration, efficiency, disturbances, and daytime dysfunction, evaluated using the Pittsburgh Sleep Quality Index (PSQI) | 6 months
  To evaluate sleep quality, latency, duration, efficiency, disturbances, and daytime dysfunction. The PSQI consists of 19 individual items, which are combined to form seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored on a 0-3 scale, and the sum of these scores yields one global score.
Overall quality of life (QOL-AD Questionnaire) | 6 months
  To gauge overall quality of life. QOL-AD is a 15-question tool used for assessing the quality of life in patients diagnosed with dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sultan Abdul Aziz Shah, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No